CLINICAL TRIAL: NCT04224038
Title: The Inspire Bio-resource Research Platform for Healthy Aging
Brief Title: The Inspire Bio-resource Research Platform for Healthy Aging INSPIRE Platform
Acronym: INSPIRE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: European Regional Development Fund (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0236
Record Dates: First submitted 2019-10-15; First posted 2020-01-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Biological Aging
Keywords: Geroscience; biological aging and identifying targetable biomarkers; The Inspire Bio-resource Research Platform for Healthy Aging; Aged 30 years-old or over; age-related chronic diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Inspire Bio-resource Research Platform for Healthy Aging — Several follow-up visits will be undertaken during the 10-year time frame of this project. Some of these visits are not regularly scheduled and will be conditioned by the remote monitoring of intrinsic capacity (IC) and the onset of other major clinical conditions. Other visits correspond to the regularly scheduled (yearly or every two years (biannual visits), depending on the outcome measures) waves of data collection.

SUMMARY:
Since aging is a systemic (not organ-specific) phenomenon, the main objective of Inspire Bio-resource Research Platform for Healthy Aging is to build a comprehensive research platform gathering biological, clinical (including imaging) and digital resources that will be explored to identify robust (set of) markers of aging, age-related diseases and IC evolution. The Inspire Platform will gather data and biospecimens from subjects of different ages (from 30 years or over - no upper limit for age) and functional capacity levels (from robust to frail to disabled) over 10 years.

DETAILED DESCRIPTION:
This is a 10-year observational study. The study will be performed in Occitania Region. Once a year, a complete data collection will be performed in the Gerontopole of Toulouse, in participants' home and health centers by the Gerontopole mobile research team, and in selected Gerontopole's collaborating centers in Occitania.

Between yearly waves of data collection, participants will have their intrinsic capacity domains monitored (with or without the help of a caregiver) each 4-month through the use of either an app developed in collaboration with World Health Organization (WHO) or a web platform; or through a phone call by a clinical/research nurse. For the first self-monitoring of IC at four months, all participants will be contacted by a research/clinical nurse by phone; this call will inform about how participants measured their capacity and/or help them to do it. After this first 4-month phone call, participants capable of correctly self-monitoring their IC through the app will no longer be systematically contacted by phone. Once IC declines are confirmed, participants will have a thorough clinical assessment and blood sampling; such information will allow us to investigate the response of markers of aging at the time declines are detected. Those needing usual care, will be followed according to WHO framework recommendations proposed for Integrated Care for Older Adults (ICOPE).

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 years-old or over;
* Both sexes
* Affiliated to a social security scheme

Exclusion Criteria:

* severe disease compromising life expectancy at 5 years;
* Deprived of their liberty by administrative or judicial decision, or under guardianship

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will be stratified per 10-year age groups, oversampling older people in order to be able to investigate major clinical events (eg, declines on IC, onset of age-related diseases)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2031-10-16 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
Data collection of key variables and biospecimens | through study completion, an average of 10 years
  The main outcome of Inspire Bio-resource Research Platform for Healthy Aging is to build a comprehensive research platform gathering biological, clinical (including imaging) and digital resources that will be explored to identify robust (set of) markers of aging, age-related diseases and intrinsic capacities (cognition, mobility, nutrition, hearing and visual capacities, psychological capacity) evolution. The Inspire Platform will gather data and biospecimens from subjects of different ages (from 30 years or over - no upper limit for age) and functional capacity levels (from robust to frail to disabled) over 10 years.

SECONDARY OUTCOMES:
Identification of (a set of) biomarkers of aging through the constitution of a comprehensive biobank comprising: blood, saliva, urine, nasopharyngeal swabbing, skin biopsies and surface samples, dental plaque, faeces, hair bulb. | through study completion, an average of 10 years
  1. Markers of aging: The identification of (a set of) markers of aging will be allowed from the constitution of a large dataset of clinical, para-clinical and digital data as well as a comprehensive biobank comprising: blood, saliva, urine, nasopharyngeal swabbing, skin material (swabbing, stripping, biopsies), dental plaque, feces, hair bulb.
  In this part of the study, we will take advantage of three complimentary approaches to look for the best markers of aging: without a priori approach (omics: transcriptomics, proteomics, lipidomics); semi a priori approach (field-specific omic. I.e. metabolism, inflammation, cell cycle, mitochondrial network…); and targeted approach (pre-identified targets).
measure intrinsic capacity domains with questionnaire in ICOPE App (developed in collaboration with W.H.O.) | through study completion, an average of 10 years
  Icope app (developed in collaboration with W.H.O.) for smartphone and tablet to measure intrinsic capacity domains. This app will be used for the remote (at-distance) evaluation and monitoring (self-monitoring, monitoring by a caregiver, or a healthcare provider) of intrinsic capacity domains; for the monitoring, we will use only the Icope Step 1. When declines are detected in the Icope Step 1, we will use the Icope Step 2 (data collected by research nurses in a home visit or at the research facility) to confirm the decline and, then, look for the causes determining such declines.
Basic and instrumental activities of daily living. | through study completion, an average of 10 years
  Basic and instrumental activities of daily living (ADL). Basic ADLs will be assessed using the 6-item (eg, bathing, feeding, dressing) Katz scale; instrumental ADLs (IADL) will be assessed using the 8-item (eg, cooking, manipulating money) Lawton scale. These variables are measured as a clinical measurement of functional ability and, thus, healthy aging in late ages, according to WHO definition.
Mini-nutritional assessment and food frequency questionnaire. | through study completion, an average of 10 years
  Mini-nutritional assessment (MNA) and food frequency questionnaire. Nutritional status will be evaluated using the MNA (see Vitality description in Icope Step 2). A short (12-item; the question on physical activity has been removed since already investigated using other assessment tools in this project) food frequency questionnaire will be used to assess dietary quality. Nutritional status and diet may affect both intrinsic capacity domains and potential biomarkers of aging.
Lifestyle questionnaires | through study completion, an average of 10 years
  . Lifestyle questionnaires:
  1. Physical activity (PA) and sedentary time: Based on the International Physical Activity Questionnaire (IPAQ) long form.
  2. Smoking: This will be evaluated by two questions: Do you currently smoke: any tobacco product? ; e-cigarettes? Responses will be anchored by the terms: daily; weekly, but not daily; less often than weekly; not at all.
  3. Alcohol consumption: This will be evaluated by a question of the food frequency questionnaire
  4. Solar exposure: Sun Protection and Exposure Habits Questionnaires
ActivPAL: objectively physical activity parameters. | through study completion, an average of 10 years
  Objectively measured physical activity (PA) and sleep parameters. This will be assessed with an activPal activity monitor. Participants will wear the activPal for one week every two-years and will bring it back personally to the research facilities. Attention will be paid for participants wearing the activity monitor always during the same season to avoid bias related to seasonal changes. PA is one of the most important behaviors for healthy aging, being associated with both intrinsic capacity domains and biomarkers. Sleep changes are often associated with aging and may affect healthy aging.
Self-reported visceral pain. | through study completion, an average of 10 years
  Visceral pain. This will be assessed with a 4-item self-reported questionnaire. This questionnaire is particularly important for investigations on biomarkers from feces.
Participant-reported outcome for cognition (CFI) | through study completion, an average of 10 years
  Patient reported outcome measures (PROM). Four PROMs, covering cognition and mobility (the two functions that largely determine disability and increased healthcare costs), the overall feeling of fatigue and social isolation. All of them are validated tools for cognition, we will use the Cognitive Function Instrument (CFI), a 14-item questionnaire with score varying from 0 to 14, higher is worse. All the other three PROMs come from the NIH-funded initiative "Patient-reported outcomes measurement information system"
Participant-reported outcome for mobility | through study completion, an average of 10 years
  Patient reported outcome measures (PROM). Four PROMs, covering cognition and mobility (the two functions that largely determine disability and increased healthcare costs), the overall feeling of fatigue and social isolation. All of them are validated tools for cognition, we will use the Cognitive Function Instrument (CFI), a 14-item questionnaire with score varying from 0 to 14, higher is worse. All the other three PROMs come from the NIH-funded initiative "Patient-reported outcomes measurement information system"
Participant-reported outcome for fatigue | through study completion, an average of 10 years
  Patient reported outcome measures (PROM). Four PROMs, covering cognition and mobility (the two functions that largely determine disability and increased healthcare costs), the overall feeling of fatigue and social isolation. All of them are validated tools for cognition, we will use the Cognitive Function Instrument (CFI), a 14-item questionnaire with score varying from 0 to 14, higher is worse. All the other three PROMs come from the NIH-funded initiative "Patient-reported outcomes measurement information system"
Participant-reported outcome for social isolation (PROMIS) | through study completion, an average of 10 years
  Patient reported outcome measures (PROM). Four PROMs, covering cognition and mobility (the two functions that largely determine disability and increased healthcare costs), the overall feeling of fatigue and social isolation. All of them are validated tools for cognition, we will use the Cognitive Function Instrument (CFI), a 14-item questionnaire with score varying from 0 to 14, higher is worse. All the other three PROMs come from the NIH-funded initiative "Patient-reported outcomes measurement information system"
Participant-reported outcome for SARQoL. | through study completion, an average of 10 years
  Patient reported outcome measures (PROM). Four PROMs, covering cognition and mobility (the two functions that largely determine disability and increased healthcare costs), the overall feeling of fatigue and social isolation. All of them are validated tools for cognition, we will use the Cognitive Function Instrument (CFI), a 14-item questionnaire with score varying from 0 to 14, higher is worse. All the other three PROMs come from the NIH-funded initiative "Patient-reported outcomes measurement information system"
Participant-reported outcome for cognition (CFI) and mobility, fatigue, and social isolation (PROMIS), and SARQoL. | through study completion, an average of 10 years
  Patient reported outcome measures (PROM). Four PROMs, covering cognition and mobility (the two functions that largely determine disability and increased healthcare costs), the overall feeling of fatigue and social isolation. All of them are validated tools for cognition, we will use the Cognitive Function Instrument (CFI), a 14-item questionnaire with score varying from 0 to 14, higher is worse. All the other three PROMs come from the NIH-funded initiative "Patient-reported outcomes measurement information system"
Oral Health Assessment Tool (OHAT). | through study completion, an average of 10 years
  Oral Health Assessment Tool (OHAT) provides a global overview of oral health. It is composed of 8 items: lips, tongue, gum-mucosa, saliva, natural teeth, prostheses, oral hygiene and pain. Each item is scored 0, 1 or 2. A score of 0 indicates the absence of degradation, a score of 2 indicates a significant presence of degradation, a score of 1 indicates that there is a remarkable modification without a significant or widespread degradation. The minimum score is 0 (satisfactory oral status) and the maximum score is 16 (degraded oral status).
Short physical performance battery and 30-sec chair rise test. | through study completion, an average of 10 years
  Short physical performance battery (SPPB) and 30-sec chair rise test. The SPPB will be evaluated. With the participants' consent, performance in the SPPB tests will be video-recorded using standard cameras placed in three different angles in the room: the images will be analyzed to look for digital markers of aging through the patterns of motor function and subsequent subjects risk-stratification. The number of chair rises within 30secwill also be assessed in a fraction of participants. These measurements provide clinical information about mobility.
The mini-mental state examination (MMSE) | through study completion, an average of 10 years
  The Mini-mental state examination (MMSE) and neuropsychological tests. The MMSE is a scale that provides total scores ranging from 0 to 30 (higher values represent better cognitive function). Besides the MMSE, in subjects less than 70 years-old the following neuropsychological tests will be used: free and total recall of the Free and Cued Selective Reminding Test, the Digit Symbol Substitution Test, score from the Wechsler Adult Intelligence Scale-Revised, and the Category Naming Test (2-minute category fluency in animals); when combined in a composite Z-score, these variables provide accurate information about participants' cognitive function.
neuropsychological tests. | through study completion, an average of 10 years
  The Mini-mental state examination (MMSE) and neuropsychological tests. The MMSE is a scale that provides total scores ranging from 0 to 30 (higher values represent better cognitive function). Besides the MMSE, in subjects less than 70 years-old the following neuropsychological tests will be used: free and total recall of the Free and Cued Selective Reminding Test, the Digit Symbol Substitution Test, score from the Wechsler Adult Intelligence Scale-Revised, and the Category Naming Test (2-minute category fluency in animals); when combined in a composite Z-score, these variables provide accurate information about participants' cognitive function.
Skin elasticity (cutometer measurement) | through study completion, an average of 10 years
  Skin elasticity (cutometer measurement). This measures the bio-mechanical properties of the skin by applying mechanical stress to the skin. The measuring principle is based on suction and elongation. A device will be used to generate a negative pressure which can vary between 20 and 500 mbar. The area of the skin to be measured is drawn into the probe opening by this pressure. The depth of skin penetration inside the probe opening is determined by an optical measurement system. The stress can be exerted at different depths of the skin: the 2mm probe solicits the skin at the superficial dermis; the 6mm probe engages the skin more deeply, at the level of the deep dermis, at the limit of the hypodermis.
Dual Energy X-ray absorptiometry | through study completion, an average of 10 years
  Whole body magnetic resonance to measure the Isokinetic muscle strength with Dual Energy X-ray absorptiometry (DEXA°
maximum oxygen consumption | through study completion, an average of 10 years
  maximum oxygen consumption (VO²max) and aerobic power (blood sampling before and after the effort).

CONTACTS AND LOCATIONS:
Overall Officials: Bruno VELLAS, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bellelli F, Raffin J, Cesari M, Guyonnet S, Furman D, Rolland Y, Vellas B, de Souto Barreto P; IHU HealthAge INSPIRE Platform Group; IHU HealthAge Open Science group. The association of pain with intrinsic capacity and the moderating role of inflammation in France: a cross-sectional analysis of the INSPIRE-T project. Lancet Healthy Longev. 2025 Dec;6(12):100798. doi: 10.1016/j.lanhl.2025.100798. Epub 2025 Dec 5. PMID 41360071